CLINICAL TRIAL: NCT03408171
Title: 19-Gauge Fine Needle Aspirate (FNA) Versus 19-Gauge Fine Needle Biopsy (FNB) Needles for Endoscopic Ultrasound Guided Liver Biopsy (EUS-LB): A Randomized Prospective Trial
Brief Title: Comparison of 19g FNA and 19g FNB Needles for EUS-LB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-0391
Record Dates: First submitted 2017-12-06; First posted 2018-01-23 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Abnormal Liver Function
Keywords: liver biopsy; endoscopic ultrasound guided liver biopsy; FNA; FNB
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 19-gauge FNA needle (Active Comparator): A 19-gauge FNA needle will be used to obtain liver tissue during an endoscopic-ultrasound guided liver biopsy. Tissue yield and diagnostic accuracy will be assessed and compared to that of the 19-gauge FNB needle.
  Interventions: Device: 19-gauge FNA needle
- 19-gauge FNB needle (Active Comparator): A 19-gauge FNB needle will be used to obtain liver tissue during an endoscopic-ultrasound guided liver biopsy. Tissue yield and diagnostic accuracy will be assessed and compared to that of the 19-gauge FNA needle.
  Interventions: Device: 19-gauge FNB needle

INTERVENTIONS:
Device: 19-gauge FNA needle — A 19-gauge FNA needle will be used to obtain liver tissue during an endoscopic-ultrasound guided liver biopsy. Tissue yield and diagnostic accuracy will be assessed and compared to that of the 19-gauge FNB needle.
  Arms: 19-gauge FNA needle
Device: 19-gauge FNB needle — A 19-gauge FNB needle will be used to obtain liver tissue during an endoscopic-ultrasound guided liver biopsy. Tissue yield and diagnostic accuracy will be assessed and compared to that of the 19-gauge FNA needle.
  Arms: 19-gauge FNB needle

SUMMARY:
Chronic liver disorders (CLD) are a major cause of morbidity and mortality for individuals in the US. Though serologic analysis will often lead to a conclusive diagnosis, liver biopsy remains an important method for helping to determine the etiology and stage of LD. Percutaneous liver biopsy (PLB), transjugular liver biopsy (TLB) and surgical liver biopsy (SLB) are alternative methods for obtaining hepatic tissue. In recent years endoscopic ultrasound guided-liver biopsy (EUS-LB) has come to the forefront as a safe and effective method for obtaining tissue in CLD. There are several studies of the safety of EUS-LB as well as the adequacy of specimens obtained in this fashion. Most studies involve a 19-g needle, therefore in this study we hope to compare the tissue yields of a 19-g fine needle biopsy (FNB) needle, in comparison to conventional 19-g fine needle aspiration (FNA) needle. We predict that 19-g FNA and 19-g FNB needle will demonstrate similar diagnostic accuracy, with less visible blood artifact. Similarly, we predict the safety to be equal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing EUS-LB
2. Platelet count > 50,000
3. International normalized ratio (INR) < 1.5
4. Age > 18 years
5. Non-pregnant patients

Exclusion Criteria:

1. Age < 18 years
2. Pregnant patients
3. Inability to obtain consent
4. Anticoagulants or anti-platelet agents use (excluding aspirin) within the last 7-10 days
5. Platelet count < 50,000
6. INR > 1.5
7. Presence of ascites
8. Known liver cirrhosis
9. Hemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Diehl, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

REFERENCES:
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Rockey DC, Bissell DM. Noninvasive measures of liver fibrosis. Hepatology. 2006 Feb;43(2 Suppl 1):S113-20. doi: 10.1002/hep.21046. PMID 16447288
- [Background] Ziol M, Handra-Luca A, Kettaneh A, Christidis C, Mal F, Kazemi F, de Ledinghen V, Marcellin P, Dhumeaux D, Trinchet JC, Beaugrand M. Noninvasive assessment of liver fibrosis by measurement of stiffness in patients with chronic hepatitis C. Hepatology. 2005 Jan;41(1):48-54. doi: 10.1002/hep.20506. PMID 15690481
- [Background] Sherlock S, Dick R, Van Leeuwen DJ. Liver biopsy today. The Royal Free Hospital experience. J Hepatol. 1985;1(1):75-85. doi: 10.1016/s0168-8278(85)80070-2. PMID 3902951
- [Background] Eisenberg E, Konopniki M, Veitsman E, Kramskay R, Gaitini D, Baruch Y. Prevalence and characteristics of pain induced by percutaneous liver biopsy. Anesth Analg. 2003 May;96(5):1392-1396. doi: 10.1213/01.ANE.0000060453.74744.17. PMID 12707140
- [Background] Firpi RJ, Soldevila-Pico C, Abdelmalek MF, Morelli G, Judah J, Nelson DR. Short recovery time after percutaneous liver biopsy: should we change our current practices? Clin Gastroenterol Hepatol. 2005 Sep;3(9):926-9. doi: 10.1016/s1542-3565(05)00294-6. PMID 16234032
- [Background] Stone MA, Mayberry JF. An audit of ultrasound guided liver biopsies: a need for evidence-based practice. Hepatogastroenterology. 1996 Mar-Apr;43(8):432-4. PMID 8714240
- [Background] McGill DB, Rakela J, Zinsmeister AR, Ott BJ. A 21-year experience with major hemorrhage after percutaneous liver biopsy. Gastroenterology. 1990 Nov;99(5):1396-400. doi: 10.1016/0016-5085(90)91167-5. PMID 2101588
- [Background] Janes CH, Lindor KD. Outcome of patients hospitalized for complications after outpatient liver biopsy. Ann Intern Med. 1993 Jan 15;118(2):96-8. doi: 10.7326/0003-4819-118-2-199301150-00003. PMID 8416324
- [Background] Huang JF, Hsieh MY, Dai CY, Hou NJ, Lee LP, Lin ZY, Chen SC, Wang LY, Hsieh MY, Chang WY, Yu ML, Chuang WL. The incidence and risks of liver biopsy in non-cirrhotic patients: An evaluation of 3806 biopsies. Gut. 2007 May;56(5):736-7. doi: 10.1136/gut.2006.115410. No abstract available. PMID 17440193
- [Background] Bravo AA, Sheth SG, Chopra S. Liver biopsy. N Engl J Med. 2001 Feb 15;344(7):495-500. doi: 10.1056/NEJM200102153440706. No abstract available. PMID 11172192
- [Background] Bull HJ, Gilmore IT, Bradley RD, Marigold JH, Thompson RP. Experience with transjugular liver biopsy. Gut. 1983 Nov;24(11):1057-60. doi: 10.1136/gut.24.11.1057. PMID 6629116
- [Background] Poniachik J, Bernstein DE, Reddy KR, Jeffers LJ, Coelho-Little ME, Civantos F, Schiff ER. The role of laparoscopy in the diagnosis of cirrhosis. Gastrointest Endosc. 1996 Jun;43(6):568-71. doi: 10.1016/s0016-5107(96)70192-x. PMID 8781934
- [Background] Denzer U, Arnoldy A, Kanzler S, Galle PR, Dienes HP, Lohse AW. Prospective randomized comparison of minilaparoscopy and percutaneous liver biopsy: diagnosis of cirrhosis and complications. J Clin Gastroenterol. 2007 Jan;41(1):103-10. doi: 10.1097/01.mcg.0000225612.86846.82. PMID 17198072
- [Background] Diehl DL, Johal AS, Khara HS, Stavropoulos SN, Al-Haddad M, Ramesh J, Varadarajulu S, Aslanian H, Gordon SR, Shieh FK, Pineda-Bonilla JJ, Dunkelberger T, Gondim DD, Chen EZ. Endoscopic ultrasound-guided liver biopsy: a multicenter experience. Endosc Int Open. 2015 Jun;3(3):E210-5. doi: 10.1055/s-0034-1391412. Epub 2015 Feb 27. PMID 26171433
- [Background] DeWitt J, LeBlanc J, McHenry L, Ciaccia D, Imperiale T, Chappo J, Cramer H, McGreevy K, Chriswell M, Sherman S. Endoscopic ultrasound-guided fine needle aspiration cytology of solid liver lesions: a large single-center experience. Am J Gastroenterol. 2003 Sep;98(9):1976-81. doi: 10.1111/j.1572-0241.2003.07638.x. PMID 14499774
- [Background] tenBerge J, Hoffman BJ, Hawes RH, Van Enckevort C, Giovannini M, Erickson RA, Catalano MF, Fogel R, Mallery S, Faigel DO, Ferrari AP, Waxman I, Palazzo L, Ben-Menachem T, Jowell PS, McGrath KM, Kowalski TE, Nguyen CC, Wassef WY, Yamao K, Chak A, Greenwald BD, Woodward TA, Vilmann P, Sabbagh L, Wallace MB. EUS-guided fine needle aspiration of the liver: indications, yield, and safety based on an international survey of 167 cases. Gastrointest Endosc. 2002 Jun;55(7):859-62. doi: 10.1067/mge.2002.124557. PMID 12024141
- [Background] Sey MS, Al-Haddad M, Imperiale TF, McGreevy K, Lin J, DeWitt JM. EUS-guided liver biopsy for parenchymal disease: a comparison of diagnostic yield between two core biopsy needles. Gastrointest Endosc. 2016 Feb;83(2):347-52. doi: 10.1016/j.gie.2015.08.012. Epub 2015 Aug 13. PMID 26278654
- [Background] Dewitt J, McGreevy K, Cummings O, Sherman S, Leblanc JK, McHenry L, Al-Haddad M, Chalasani N. Initial experience with EUS-guided Tru-cut biopsy of benign liver disease. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):535-42. doi: 10.1016/j.gie.2008.09.056. PMID 19231495
- [Background] Gor N, Salem SB, Jakate S, Patel R, Shah N, Patil A. Histological adequacy of EUS-guided liver biopsy when using a 19-gauge non-Tru-Cut FNA needle. Gastrointest Endosc. 2014 Jan;79(1):170-2. doi: 10.1016/j.gie.2013.06.031. Epub 2013 Jul 31. No abstract available. PMID 23916397
- [Background] Stavropoulos SN, Im GY, Jlayer Z, Harris MD, Pitea TC, Turi GK, Malet PF, Friedel DM, Grendell JH. High yield of same-session EUS-guided liver biopsy by 19-gauge FNA needle in patients undergoing EUS to exclude biliary obstruction. Gastrointest Endosc. 2012 Feb;75(2):310-8. doi: 10.1016/j.gie.2011.09.043. PMID 22248599
- [Background] Colloredo G, Guido M, Sonzogni A, Leandro G. Impact of liver biopsy size on histological evaluation of chronic viral hepatitis: the smaller the sample, the milder the disease. J Hepatol. 2003 Aug;39(2):239-44. doi: 10.1016/s0168-8278(03)00191-0. PMID 12873821
- [Background] Crawford AR, Lin XZ, Crawford JM. The normal adult human liver biopsy: a quantitative reference standard. Hepatology. 1998 Aug;28(2):323-31. doi: 10.1002/hep.510280206. PMID 9695993
- [Background] Rocken C, Meier H, Klauck S, Wolff S, Malfertheiner P, Roessner A. Large-needle biopsy versus thin-needle biopsy in diagnostic pathology of liver diseases. Liver. 2001 Dec;21(6):391-7. doi: 10.1034/j.1600-0676.2001.210605.x. PMID 11903883
- [Background] Bhatia V, Hijioka S, Hara K, Mizuno N, Imaoka H, Yamao K. Endoscopic ultrasound description of liver segmentation and anatomy. Dig Endosc. 2014 May;26(3):482-90. doi: 10.1111/den.12216. Epub 2013 Dec 19. PMID 24355092
- [Background] ASGE Standards of Practice Committee; Early DS, Acosta RD, Chandrasekhara V, Chathadi KV, Decker GA, Evans JA, Fanelli RD, Fisher DA, Fonkalsrud L, Hwang JH, Jue TL, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf RN, Shergill AK, Cash BD. Adverse events associated with EUS and EUS with FNA. Gastrointest Endosc. 2013 Jun;77(6):839-43. doi: 10.1016/j.gie.2013.02.018. No abstract available. PMID 23684089
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: Years] | 51 [28 to 67] | 49 [27 to 69] | 51 [27 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  White (Non-hispanic) | 18 | 16 | 34
  White (Hispanic) | 1 | 3 | 4
  Afroamerican | 0 | 1 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Pre-processing Length of the Longest Piece (LLP)
Description: Pre-processing Length of the longest piece (LLP) measured in centimeter
Time Frame: up to 5 days
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
centimeter | 1.47 (0.46) | 2.09 (0.41)

2. Secondary Outcome: Post-processing Length of the Longest Piece (LLP)
Description: Post-processing Length of the longest piece (LLP) measured in centimeter
Time Frame: 3-5 days
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
centimeter | 1.05 (0.42) | 1.78 (0.66)

3. Secondary Outcome: Number of Participants With LLP Pre-processing Length Less Than 2 cm or Greater Than 2 cm
Description: Pre-processing Length of the longest piece (LLP) subgroups:
  < 2 cm > 2cm
Time Frame: 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
Participants
  < 2 cm | 17 | 10
  > 2 cm | 3 | 10

4. Secondary Outcome: Pre-processing Aggregate Specimen Length (ASL)
Description: Pre-processing Aggregate specimen length (ASL) measured in centimeter
Time Frame: 3-5 days
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
centimeter | 10.89 (4.38) | 15.78 (5.19)

5. Secondary Outcome: Post-processing Aggregate Specimen Length (ASL)
Description: Post-processing Aggregate specimen length (ASL) measured in centimeter
Time Frame: 3-5 days
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
centimeter | 11.4 (5.55) | 15.32 (5.24)

6. Secondary Outcome: Portal Triads Number (Mean)
Description: Number of portal triads (PT) in the specimen.
Time Frame: 3-5 days
Measure: Mean (Standard Deviation); unit: Portal Triads
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
Portal Triads | 18.1 (9.3) | 42.6 (25)

7. Secondary Outcome: Portal Triads Quantity (Median)
Description: Number of portal triads (PT) in the specimen.
Time Frame: 3-5 days
Measure: Median (Full Range); unit: Complete number of portal triads
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
Complete number of portal triads | 16.5 [6 to 38] | 38 [0 to 81]

8. Secondary Outcome: Number of Participants With Fewer Than 11 Portal Triads or More Than 11 Portal Triads
Description: Portal triads groups, n (%) < 11 Portal triads > 11 Portal triads
Time Frame: 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
Participants
  < 11 Portal triads | 6 | 2
  > Portal triads | 14 | 18

9. Secondary Outcome: No. of Fragments > 9 mm, Mean (SD)
Description: No. of fragments > 9 mm, mean (SD) Pre-processing Post-processing
Time Frame: 3-5 days
Measure: Mean (Standard Deviation); unit: Number of Fragments
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
Number of Fragments
  Pre-processing | 3.5 (2.4) | 7.7 (3.7)
  Post-processing | 1.1 (1) | 4.8 (3.6)

10. Secondary Outcome: Specimen Quality for Histologic Diagnosis
Description: Number of cases for which a histologic diagnosis could be made based upon the amount of tissue obtained with the needle.
Time Frame: 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

11. Secondary Outcome: Length of Longest Piece
Time Frame: Number Analyzed
Measure: Median (Full Range); unit: mm
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
Number analyzed (Participants) | 20 | 20
mm | 32.3 [21.6 to 49.5] | 30.2 [21.6 to 50]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | 19-gauge FNA Needle | 19-gauge FNB Needle
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 19-gauge FNA Needle (N=20) | 19-gauge FNB Needle (N=20)
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Headache (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Research was completed at a high-volume center; therefore, our outcomes may not be fully applicable to small practices.

Learning curve to achieving best possible tissue samples with EUS-LB, which appears to be between 10 and 20 procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03408171/Prot_SAP_000.pdf